CLINICAL TRIAL: NCT01460277
Title: Τhe Effectiveness of Hydrotherapy Exercises on the Rehabilitation of Hemiplegic Patients
Acronym: hydro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Avraam Ploumis, Assistant Professor of PMR, Orthopaedic Spine Surgeon, University of Ioannina
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 275/2011
Record Dates: First submitted 2011-10-22; First posted 2011-10-26 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Hemiplegics
Keywords: hemiplegic; balance; hydrotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Hydrokinesiotherapy (Experimental): A 6-week water-based exercise program that focused on balance and weight bearing exercises (3 days a week for 1 hour a session)
  Interventions: Procedure: Hydrokinesiotherapy Intervention
- Conventional exercise intervention (Active Comparator): A 6-week land-based exercise program that focused on balance and weight bearing exercises (3 days a week for 1 hour a session)
  Interventions: Procedure: Land-based exercise intervention

INTERVENTIONS:
Procedure: Hydrokinesiotherapy Intervention — The hydrotherapy exercise intervention consisted of 5 minutes of warm-up, 10 minutes of lower-extremity stretching exercises, 10 minutes of lower-extremity strengthening exercises, 20 minutes balance and gait training (water walking, running, side stepping), 5 minutes of a light cool down (marching on the spot), and 10 minutes of gentle stretching in the water.
  Arms: Hydrokinesiotherapy
Procedure: Land-based exercise intervention — The conventional exercise intervention used no water-based exercises but land-based exercises. The exercise program consisted of 5 minutes of warm-up, 10 minutes of lower-extremity stretching exercises, 10 minutes of lower-extremity strengthening exercises, 20 minutes balance and gait training (walking, side stepping), 5 minutes of a light cool down, and 10 minutes of gentle stretching out of the water.
  Arms: Conventional exercise intervention

SUMMARY:
The purpose of this current prospective study is to assess and compare the effects of a hydrotherapy exercise programme against a conventional land-based exercise programme in individuals with hemiplegia. Both exercise interventions aim at improving posture, balance and weight-bearing capability. Patients were randomized to the hydrotherapy or conventional therapy groups according to balance function (Berg Balance Scale score) and age (age<59 and >60 years). The physical examination consisted of (1) a lower-limb motor function recovery of the paretic side score according to the 6-stage Brunnstrom scale, (2) the hemiplegic limb strength measured by the Motricity Index, (3) the strength of ankle dorsiflexors and plantarflexors by manual muscle testing, (4) the spasticity of the ankle score by Modified Ashworth Scale, (5) the trunk function through the Trunk Control Test, (6) the postural control assessed by Postural Assessment Scale for Stroke Patients and (7) the functional status measured with the Functional Independence Measure. Postural sway was evaluated with a pressure platform by using the variables of center of pressure (COP) displacements in the mediolateral (ML) and anteroposterior (AP) directions. The results will be collected and evaluated using statistical programme SPSS.

ELIGIBILITY:
Inclusion Criteria:

* hemiplegia or hemiparesis after stroke or traumatic brain injury
* at least 6 months post-stroke from a single cerebrovascular accident
* independent in walking (with or without assistive device)
* clinical stable

Exclusion Criteria:

* unstable cardiac conditions
* epilepsy
* urinary or faecal incontinence
* open wounds
* significant musculoskeletal problems in lower extremities from conditions other than stroke
* Alzheimer
* Parkinson's disease
* polyneuropathy
* vestibular disorders
* current participation in an exercise program

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change of postural and sitting balance at six weeks | At the time of admittance to the rehabilitation department (at baseline) and after six weeks
  Postural balance and weight-bearing ability measured by vertical ground reaction force during standing, sitting and four standing tasks (rising from a chair and weight-shifting forward, backward and laterally)

SECONDARY OUTCOMES:
Change of balance at six weeks | At the time of admittance to the rehabilitation department (at baseline) and after six weeks
  Berg Balance Score
Change of spasticity at six weeks | At the time of admittance to the rehabilitation department (at baseline) and after six weeks
  with ashworth test
Change of leg's strength at 6 weeks | At the time of admittance to the rehabilitation department (at baseline) and after six weeks
  6-stages Brunnstrom scale
Change of trunk control at 6 weeks | At the time of admittance to the rehabilitation department (at baseline) and after six weeks
  Trunk Control Test (TCT)
Change of function at 6 weeks | At the time of admittance to the rehabilitation department (at baseline) and after six weeks
  Functional Indepedence Measure (FIM)
Change of leg's motion at 6 weeks | At the time of admittance to the rehabilitation department (at baseline) and after six weeks
  Motricity Index
Change of posture at 6 weeks | At the time of admittance to the rehabilitation department (at baseline) and after six weeks
  Postural Assessment Scale for Stroke Patient (PASS)

CONTACTS AND LOCATIONS:
Overall Officials: Avraam Ploumis, Principal Investigator — University Hospital, Ioannina
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece

REFERENCES:
- [Derived] Iatridou G, Stergiou AN, Varvarousis DN, Theodorou A, Doulgeri S, Pelidou HS, Dimakopoulos G, Ploumis A. Comparative Study Between Aquatic Therapy and Land-Based Exercises in Hemiplegic Patients After Stroke: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2025 Apr 1;104(4):305-311. doi: 10.1097/PHM.0000000000002589. Epub 2024 Jul 2. PMID 38954645